CLINICAL TRIAL: NCT01272180
Title: Phase 2, Observer Blinded, Controlled, Randomized Multi-Center Study in Adolescents and Young Adults to Evaluate Safety and Immunogenicity of Two Different rMenB With OMV + MenACWY Combination Vaccination Formulations
Brief Title: Safety and Immunogenicity of Different Meningitis Vaccine Formulations in Adolescents and Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V102_03; 2010-023523-23 (EudraCT Number)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2019-03

CONDITIONS: Invasive Meningococcal Disease
Keywords: Safety; Immunogenicity; Vaccine; Meningococcal; Seroresponse

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- ABCWY+OMV (Experimental): Subjects in this group received two doses of "Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine" plus Outer Membrane Vesicles (OMV) administered two months apart.
  Interventions: Biological: Meningococcal (groups A, C, W, Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine + OMV.
- ABCWY+qOMV (Experimental): Subjects in this group received two doses of "Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine" plus one quarter dose of Outer Membrane Vesicles (qOMV) administered two months apart.
  Interventions: Biological: Meningococcal (groups A, C, W, Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine + qOMV.
- rMenB+OMV (Active Comparator): Subjects in this group received two doses of "Meningococcal (group B) multicomponent recombinant adsorbed vaccine",administered two months apart.
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine plus OMV.
- MenACWY (Active Comparator): Subjects in this group received a dose of placebo followed by one dose of "Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine" administered two months later.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine.

INTERVENTIONS:
Biological: Meningococcal (groups A, C, W, Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine + OMV. — Two injections of a combined vaccine formulation, Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine plus OMV.
  Arms: ABCWY+OMV
Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine plus OMV. — Two injections of Meningococcal (group B) multicomponent recombinant adsorbed vaccine plus OMV.
  Arms: rMenB+OMV
Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine. — One injection of saline solution placebo and one of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine.
  Arms: MenACWY
Biological: Meningococcal (groups A, C, W, Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine + qOMV. — Two injections of a combined vaccine formulation, Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine plus a quarter dose of OMV.
  Arms: ABCWY+qOMV

SUMMARY:
This study will evaluate the safety and immunogenicity of combination vaccines as compared to the reference vaccines

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents aged 10 through 25 years of age inclusive at the time of enrollment.

Exclusion Criteria:

* History of any meningococcal vaccine administration;
* Current or previous, confirmed or suspected disease caused by N. meningitidis;
* Pregnant or nursing (breastfeeding) mothers;
* Females of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study;
* Any serious, chronic, or progressive disease;
* Known or suspected impairment/alteration of the immune system;
* Receipt of blood, blood products and/or plasma derivatives, or a parenteral immunoglobulin preparation within the previous 90 days;
* History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 484 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (13):
- United States (8):
  - Alabama Clinical Therapeutics, 806 St. Vincent's Drive, Suite 615, Birmingham, Alabama
  - Madera Family Medical Group,1111 West 4th Street, Madera, California
  - Center for Clinical Trials LLC, 16660 Paramount Blvd, Suite 301, Paramount, California
  - Kentucky Pediatric/Adult Research, 201 south 5th street, Bardstown, Kentucky
  - Bluegrass Clinical Research Inc.5512 Bardstown Road, Suite 2, Louisville, Kentucky
  - Ohio Pediatric Research Association, 7371 Brandt Pike, Suite C, Huber Heights, Ohio
  - Ohio Pediatric Research Association, 1775 Delco Park Drive, Kettering, Ohio
  - Focus Research Group,201 Signature Place, Lebanon, Tennessee
- Poland (5):
  - Specjalistyczna Przychodnia Lekarska Internistyczno-Pediatryczna,,Juniperus"s.c, ul.Kościuszki 41, Izabelin (Warszawa)
  - NZOZ HIPOKRATES II.sp.zo.o, ul.Pachonskiego 12, Krakow
  - NZOZ PRAKTIMED Sp.zo.o, ul.Strzelców 15, Krakow
  - Klinika Pediatrii Centrum Medycznego Kształcenia PodyplomowegoSzpital Bielański, ul. Cegłowska 80, Warsaw
  - Katedra i Klinika Pediatrii i Chorób Infekcyjnych, ul.O.Bujwida 44, Wroclaw

REFERENCES:
- [Derived] Szenborn L, Block SL, Jackowska T, Konior R, D'Agostino D, Smolenov I, Toneatto D, Welsch JA. Immune Responses to Booster Vaccination With Meningococcal ABCWY Vaccine After Primary Vaccination With Either Investigational or Licensed Vaccines: A Phase 2 Randomized Study. Pediatr Infect Dis J. 2018 May;37(5):475-482. doi: 10.1097/INF.0000000000001896. PMID 29329168

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- ABCWY+OMV: Subjects in this group received two doses of ABCWY+OMV combination vaccine, administered two months apart.
- ABCWY+qOMV: Subjects in this group received two doses of ABCWY+qOMV combination vaccine, administered two months apart.
- rMenB +OMV: Subjects in this group received two doses of rMenB + OMV vaccine,administered two months apart.
- ACWY: Subjects in this group received one dose of placebo followed by one dose of MenACWY vaccine two months later.
Period: Overall Study
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB +OMV | ACWY
Started | 120 | 121 | 122 | 121
Completed | 103 | 100 | 109 | 107
Not Completed | 17 | 21 | 13 | 14
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 6 | 3 | 2
Not completed — Lost to Follow-up | 15 | 14 | 8 | 10
Not completed — Inappropriate enrollment | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Anaysis was done on the All Enrolled Population, ie, all subjects who signed an informed consent/assent, undergone screening procedure(s) and were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB +OMV | ACWY | Total
Number analyzed (Participants) | 120 | 121 | 122 | 121 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (4.7) | 15.1 (4.9) | 15.3 (4.9) | 15.0 (5.1) | 15.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 68 | 60 | 64 | 253
  Male | 59 | 53 | 62 | 57 | 231

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With a Seroresponse Against N.Meningitidis Serogroups A,C,W-135,Y, After Receiving Different Formulations of MenABCWY Combination Vaccine.
Description: Non-inferiority of immune response of two doses of two different formulations of MenABCWY vaccine to a single dose of MenACWY vaccine as measured by the percentage of subjects with hSBA seroresponse against N.meningitidis serogroups A,C,W and Y.
  Seroresponse is defined as:
  1. For subjects with a pre-vaccination hSBA titer < 1:4, a post-vaccination hSBA titer ≥ 1:8;
  2. For subjects with a pre-vaccination hSBA titer ≥ 1:4, an increase in hSBA titer of at least four times the prevaccination titer.
  Functional bactericidal antibodies directed against serogroups A,C,W,Y meningococci were measured with a serum bactericidal activity assay using human serum as the source of exogenous complement (hSBA).
Time Frame: One month after the second vaccination (Day 91)
Population: Analysis was done on the per protocol population, immunogenicity, i.e subjects who received correct vaccines in both the visits; provided evaluable serum sample pre and post vaccination with assay results available for at least one serogroup and/or strain and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ABCWY+OMV | ABCWY+qOMV | ACWY
Number analyzed (Participants) | 88 | 84 | 76
Percentages of subjects
  Men A: number analyzed (Participants) | 88 | 83 | 75
  Men A | 90 [81 to 95] | 92 [83 to 97] | 73 [62 to 83]
  Men C: number analyzed (Participants) | 86 | 84 | 76
  Men C | 95 [89 to 99] | 93 [85 to 97] | 63 [51 to 74]
  Men W-135: number analyzed (Participants) | 75 | 73 | 60
  Men W-135 | 80 [69 to 88] | 84 [73 to 91] | 65 [52 to 77]
  Men Y: number analyzed (Participants) | 65 | 70 | 59
  Men Y | 92 [83 to 97] | 90 [80 to 96] | 75 [62 to 85]
Statistical Analysis 1: Comparison: ABCWY+OMV vs ACWY; Non-inferiority of seroresponse against N.meningitidis serogroup A of two doses of MenABCWY combination vaccine to that of one dose of MenACWY vaccine; Test type: Non-Inferiority or Equivalence — The immune response of ABCWY+OMV group was considered to be non-inferior to that of ACWY group if the lower limit of the two-sided 95% confidence interval on the difference between groups in percentage of subjects with seroresponse is greater than -10% for each of A, C, W-135and Y serogroups, at 30 days after the last vaccination; Group Difference % (ABCWY+OMV - ACWY) = 16, 95% CI 2-sided [5 to 29]
Statistical Analysis 2: Comparison: ABCWY+OMV vs ACWY; Non-inferiority of seroresponse against N.meningitidis serogroup C of two doses of ABCWY+OMV combination vaccine to that of one dose of MenACWY vaccine; Test type: Non-Inferiority or Equivalence — The immune response of ABCWY+OMV group was considered to be non-inferior to that of ACWY group if the lower limit of the two-sided 95% confidence interval on the difference between MenABCWY and MenACWY groups in percentage of subjects with seroresponse is greater than -10% for each of A, C, W-135and Y serogroups, at 30 days after the last vaccination; Group Difference % (ABCWY+OMV - ACWY) = 32, 95% CI 2-sided [21 to 44]
Statistical Analysis 3: Comparison: ABCWY+OMV vs ACWY; Non-inferiority of seroresponse against N.meningitidis serogroup W-135 of two doses of ABCWY+OMV combination vaccine to that of one dose of MenACWY vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Group Difference % (ABCWY+OMV - ACWY) = 15, 95% CI 2-sided [0 to 30]
Statistical Analysis 4: Comparison: ABCWY+OMV vs ACWY; Non-inferiority of seroresponse against N.meningitidis serogroup Y of two doses MenABCWY combination vaccine to that of one dose of MenACWY vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Group Difference % (ABCWY+OMV - ACWY) = 18, 95% CI 2-sided [5 to 31]
Statistical Analysis 5: Comparison: ABCWY+qOMV vs ACWY; Non-inferiority of seroresponse against N.meningitidis serogroup A of two doses of MenABCWY+qOMV combination vaccine to that of one dose of MenACWY vaccine; Test type: Non-Inferiority or Equivalence — The immune response of MenABCWY+qOMV group was considered to be non-inferior to that of ACWY group if the lower limit of the two-sided 95% confidence interval on the difference between groups in percentage of subjects with seroresponse is greater than -10% for each of A, C, W-135and Y serogroups, at 30 days after the last vaccination; Group Difference % (ABCWY+qOMV - ACWY) = 18, 95% CI 2-sided [7 to 30]
Statistical Analysis 6: Comparison: ABCWY+qOMV vs ACWY; Non-inferiority of seroresponse against N.meningitidis serogroup C of two doses of MenABCWY+qOMV combination vaccine to that of one dose of MenACWY vaccine; Test type: Non-Inferiority or Equivalence — The immune response of MenABCWY+qOMV group was considered to be non-inferior to that of MenACWY group if the lower limit of the two-sided 95% confidence interval on the difference between groups in percentage of subjects with seroresponse is greater than -10% for each of A, C, W-135and Y serogroups, at 30 days after the last vaccination; Group Difference % (ABCWY+qOMV - ACWY) = 30, 95% CI 2-sided [18 to 42]
Statistical Analysis 7: Comparison: ABCWY+qOMV vs ACWY; Non-inferiority of seroresponse against N.meningitidis serogroup W-135 of two doses of MenABCWY+qOMV combination vaccine to that of one dose of MenACWY vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 6]; Group Difference % (ABCWY+qOMV - ACWY) = 19, 95% CI 2-sided [4 to 33]
Statistical Analysis 8: Comparison: ABCWY+qOMV vs ACWY; Non-inferiority of seroresponse against N.meningitidis serogroup Y of two doses of MenABCWY+qOMV combination vaccine to that of one dose of MenACWY vaccine; Test type: Non-Inferiority or Equivalence — The immune response of MenABCWY+qOMV group was considered to be non-inferior to that of MenACWY group if the lower limit of the two-sided 95% confidence interval on the difference between groups in percentage of subjects with seroresponse is greater than -10% for each of A, C, W-135and Y serogroups, at 30 days; Group Difference % (ABCWY+qOMV - ACWY) = 15, 95% CI 2-sided [3 to 29]

2. Primary Outcome: Desirability Index for Each Vaccine Group, Based on Immunogenicity and Reactogenicity Parameters.
Description: The overall desirability index (DI) used to identify the optimal formulation of the combination vaccine was based on immunogenicity and reactogenicity parameters (on a scale of 0 to 1, with 0 for an undesirable response and 1 for a highly desirable response) as follows: Between-group ratios of hSBA GMTs were calculated, adjusted for prevaccination titer and center, against serogroups A, C, W, and Y (ABCWY+OMV group or ABCWY+qOMV group vs. Placebo/ACWY group) and against the 4 serogroup B test strains (ABCWY+OMV group or ABCWY+qOMV group vs. rMenB+OMV group). Reactogenicity was measured by the percentage of doses associated with severe local and systemic solicited AEs within 3 days following vaccination. Each immunogenicity and reactogenicity endpoint was assigned its own DI based on predefined desirability functions. The overall DI was calculated using the weighted geometric mean of the DI values of each of the ten parameters to derive an overall DI for each formulation.
Time Frame: One month after the second vaccination (Day 91)
Population: Analysis was done on the Per Protocol Set - desirability, ie, all subjects who :
  correctly received the vaccine at Visit 1 and Visit 2, provided evaluable serum samples pre- (Visit 1) and post-vaccination (Visit 3), provided post-vaccination solicited adverse event data an had no major protocol violation as defined prior to unblinding.
Measure: Number; unit: Desirability index
Arm/Group | ABCWY+OMV | ABCWY+qOMV
Number analyzed (Participants) | 86 | 82
Desirability index | 0.306 | 0.325

3. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 Against N.Meningitidis Serogroups A,C,W-135 and Y, After Vaccination With Different Formulations of MenABCWY Combination Vaccine.
Description: Percentages of subjects with hSBA titers ≥ 1:8 against N.meningitidis serogroups A,C,W-135 and Y, after two doses of either ABCWY+OMV or ABCWY+qOMV combination vaccine or one dose of MenACWY vaccine.
Time Frame: Day 1 and one month after second vaccination (Day 91)
Population: Analysis was done on the per protocol population, immunogenicity.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ABCWY+OMV | ABCWY+qOMV | ACWY
Number analyzed (Participants) | 90 | 85 | 76
Percentages of subjects
  Men A (Day 1) | 8 [3 to 15] | 6 [2 to 13] | 1 [0.033 to 7]
  Men A (Day 91): number analyzed (Participants) | 88 | 83 | 75
  Men A (Day 91) | 93 [86 to 97] | 95 [88 to 99] | 73 [62 to 83]
  Men C (Day 1): number analyzed (Participants) | 88 | 85 | 76
  Men C (Day 1) | 35 [25 to 46] | 35 [25 to 46] | 32 [21 to 43]
  Men C (Day 91): number analyzed (Participants) | 86 | 84 | 76
  Men C (Day 91) | 99 [94 to 100] | 100 [96 to 100] | 83 [73 to 91]
  Men W-135 (Day 1): number analyzed (Participants) | 86 | 79 | 68
  Men W-135 (Day 1) | 66 [55 to 76] | 58 [47 to 69] | 51 [39 to 64]
  Men W-135 (Day 91): number analyzed (Participants) | 77 | 75 | 65
  Men W-135 (Day 91) | 100 [95 to 100] | 100 [95 to 100] | 89 [79 to 96]
  Men Y (Day 1): number analyzed (Participants) | 89 | 85 | 74
  Men Y (Day 1) | 18 [11 to 28] | 15 [8 to 25] | 8 [3 to 17]
  Men Y (Day 91): number analyzed (Participants) | 65 | 70 | 60
  Men Y (Day 91) | 97 [89 to 100] | 97 [90 to 100] | 82 [70 to 90]

4. Secondary Outcome: The hSBA GMTs Against N.Meningitidis Serogroups A,C,W-135 and Y, After Vaccination With Different Formulations of MenABCWY Combination Vaccine.
Description: The hSBA GMTs against N.meningitidis serogroups A,C,W-135 and Y, after two doses of either ABCWY+OMV or ABCWY+qOMV combination vaccine, or one dose of MenACWY vaccine.
Time Frame: Day 1 and one month after the second vaccination (Day 91)
Population: Analysis was done on the per protocol population, immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY+OMV | ABCWY+qOMV | ACWY
Number analyzed (Participants) | 90 | 85 | 76
Titers
  Men A (Day 1) | 1.57 [1.28 to 1.92] | 1.32 [1.07 to 1.63] | 1.33 [1.08 to 1.65]
  Men A (Day 91): number analyzed (Participants) | 88 | 83 | 75
  Men A (Day 91) | 71 [49 to 102] | 77 [53 to 111] | 45 [31 to 65]
  Men C (Day 1): number analyzed (Participants) | 88 | 85 | 76
  Men C (Day 1) | 4.15 [3.02 to 5.69] | 3.72 [2.69 to 5.12] | 3.93 [2.84 to 5.45]
  Men C (Day 91): number analyzed (Participants) | 86 | 84 | 76
  Men C (Day 91) | 214 [148 to 309] | 187 [129 to 272] | 55 [38 to 80]
  Men W-135 (Day 1): number analyzed (Participants) | 86 | 79 | 68
  Men W-135 (Day 1) | 14 [8.88 to 22] | 10 [6.45 to 16] | 6.58 [4.11 to 11]
  Men W-135 (Day 91): number analyzed (Participants) | 77 | 75 | 65
  Men W-135 (Day 91) | 239 [178 to 322] | 288 [214 to 389] | 65 [48 to 90]
  Men Y (Day 1): number analyzed (Participants) | 89 | 85 | 74
  Men Y (Day 1) | 2.01 [1.52 to 2.66] | 1.91 [1.43 to 2.53] | 1.52 [1.14 to 2.04]
  Men Y (Day 91): number analyzed (Participants) | 65 | 70 | 60
  Men Y (Day 91) | 149 [95 to 234] | 129 [83 to 201] | 46 [29 to 72]

5. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:5 and ≥ 1:8 Against N.Meningitidis Serogroup B, After Vaccination With Different Formulations of MenABCWY Combination Vaccine.
Description: The percentages of subjects with hSBA titers ≥ 1:5 and ≥ 1:8 against four different strains of N.meningitidis serogroup B, after two doses of ABCWY+OMV, ABCWY+qOMV or rMenB+OMV vaccine.
Time Frame: Day 1 and one month after the second vaccination (Day 91)
Population: Analysis was done on the per-protocol population, immunogenicity
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- rMenB +OMV: Subjects in this group received two doses of rMenB+OMV vaccine, administered two months apart.
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB +OMV
Number analyzed (Participants) | 90 | 85 | 92
Percentages of subjects
  M14459 (Day 1; hSBA ≥1:5) | 9 [4 to 17] | 4 [1 to 10] | 5 [2 to 12]
  M14459 (Day 91; hSBA ≥1:5): number analyzed (Participants) | 89 | 85 | 92
  M14459 (Day 91; hSBA ≥1:5) | 64 [53 to 74] | 71 [60 to 80] | 82 [72 to 89]
  M01-0240364 (Day 1; hSBA ≥1:5): number analyzed (Participants) | 90 | 84 | 91
  M01-0240364 (Day 1; hSBA ≥1:5) | 3 [1 to 9] | 14 [8 to 24] | 4 [1 to 11]
  M01-0240364 (Day 91; hSBA ≥1:5): number analyzed (Participants) | 86 | 84 | 90
  M01-0240364 (Day 91; hSBA ≥1:5) | 80 [70 to 88] | 80 [70 to 88] | 93 [86 to 98]
  NZ 98/254 (Day 1; hSBA ≥1:5): number analyzed (Participants) | 89 | 85 | 92
  NZ 98/254 (Day 1; hSBA ≥1:5) | 3 [1 to 10] | 1 [0.03 to 6] | 3 [1 to 9]

6. Secondary Outcome: Percentages of Subjects With at Least 4-fold Increase in hSBA Titers Against N.Meningitidis Serogroup B, After Vaccination With Different Formulations of MenABCWY Combination Vaccine.
Description: The percentages of subjects with at least 4-fold increase in hSBA titers against four different strains of N.meningitidis serogroup B, after two doses of ABCWY+OMV, ABCWY+qOMV or rMenB+OMV vaccine.
  4-fold increase is defined as follows;
  for subjects with a prevaccination hSBA < 1:2, a postvaccination hSBA ≥ 1:8, for subjects with a prevaccination hSBA ≥ 1:2, at least a 4-fold increase.
Time Frame: One month after the second vaccination (Day 91)
Population: Analysis was done on the per-protocol population, immunogenicity.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- rMenB+OMV: Subjects in this group received two doses of rMenB+OMV vaccine, administered two months apart.
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB+OMV
Number analyzed (Participants) | 89 | 85 | 92
Percentages of subjects
  M14459 | 56 [45 to 67] | 62 [51 to 73] | 75 [65 to 83]
  M01-0240364: number analyzed (Participants) | 86 | 83 | 89
  M01-0240364 | 79 [69 to 87] | 70 [59 to 79] | 88 [79 to 94]
  NZ98/254: number analyzed (Participants) | 88 | 84 | 92
  NZ98/254 | 47 [36 to 58] | 48 [37 to 59] | 76 [66 to 84]
  M07-0241084: number analyzed (Participants) | 87 | 84 | 92
  M07-0241084 | 28 [19 to 38] | 25 [16 to 36] | 42 [32 to 53]

7. Secondary Outcome: The hSBA GMTs Against N.Meningitidis serogroupB, After Vaccination With Different Formulations of MenABCWY Combination Vaccine.
Description: The hSBA GMTs against N.meningitidis serogroup B after two doses of ABCWY+OMV, ABCWY+qOMV or rMenB+OMV vaccine.
Time Frame: Day 1 and one month after the second vaccination (Day 91)
Population: Analysis was done on the per-protocol population, immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- rMenB +OMV: Subjects in this group received two doses of rMenB + OMV vaccine, administered two months apart.
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB +OMV
Number analyzed (Participants) | 90 | 85 | 92
Titers
  M14459 (Day 1) | 1.32 [1.09 to 1.59] | 1.15 [0.95 to 1.4] | 1.26 [1.04 to 1.53]
  M14459 (Day 91): number analyzed (Participants) | 89 | 85 | 92
  M14459 (Day 91) | 9.24 [6.19 to 14] | 11 [7.51 to 17] | 17 [11 to 25]
  M01-0240364 (Day 1): number analyzed (Participants) | 90 | 84 | 91
  M01-0240364 (Day 1) | 1.08 [0.82 to 1.42] | 1.72 [1.29 to 2.28] | 1.14 [0.86 to 1.51]
  M01-0240364 (Day 91): number analyzed (Participants) | 86 | 84 | 90
  M01-0240364 (Day 91) | 55 [33 to 93] | 48 [28 to 83] | 118 [69 to 202]
  NZ 98/254 (Day 1): number analyzed (Participants) | 89 | 85 | 92
  NZ 98/254 (Day 1) | 1.2 [1.03 to 1.39] | 1.1 [0.94 to 1.28] | 1.21 [1.04 to 1.42]
  NZ 98/254 (Day 91): number analyzed (Participants) | 89 | 84 | 92
  NZ 98/254 (Day 91) | 8.68 [5.91 to 13] | 7.88 [5.3 to 12] | 19 [13 to 27]
  M07-0241084 (Day 1): number analyzed (Participants) | 89 | 84 | 92
  M07-0241084 (Day 1) | 2.55 [1.86 to 3.49] | 2.45 [1.76 to 3.4] | 2.13 [1.54 to 2.94]
  M07-0241084 (Day 91): number analyzed (Participants) | 88 | 85 | 92
  M07-0241084 (Day 91) | 7.24 [5.4 to 9.71] | 6.26 [4.63 to 8.46] | 12 [8.83 to 16]

8. Secondary Outcome: The Geometric Mean Ratio of Post vs Pre Vaccination GMTs Against N.Meningitidis Serogroup B, After Vaccination With Different Formulations of MenABCWY Combination Vaccine.
Description: The geometric mean ratio (GMR) of post vaccination versus pre vaccination GMTs against N.meningitidis serogroup B after two doses of ABCWY+OMV, ABCWY+qOMV or rMenB+OMV vaccine.
Time Frame: One month after the second vaccination/prevaccination (Day 91/day 1)
Population: Analysis was done on the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB+OMV
Number analyzed (Participants) | 89 | 85 | 92
Ratio
  M14459 | 7.32 [4.89 to 11] | 9.41 [6.19 to 14] | 14 [9.01 to 21]
  M01-0240364: number analyzed (Participants) | 86 | 83 | 89
  M01-0240364 | 48 [27 to 83] | 30 [17 to 54] | 98 [56 to 173]
  NZ 98/254: number analyzed (Participants) | 88 | 84 | 92
  NZ 98/254 | 7.44 [5.06 to 11] | 6.91 [4.64 to 10] | 16 [11 to 23]
  M07-0241084: number analyzed (Participants) | 87 | 84 | 92
  M07-0241084 | 2.94 [2.15 to 4.02] | 2.59 [1.88 to 3.58] | 5.16 [3.76 to 7.08]

9. Secondary Outcome: The Number of Subjects Reporting Solicited Adverse Events After Receiving Any Vaccination in This Study.
Description: The number of subjects reporting solicited local and systemic adverse events and other indicators of reactogenicity after vaccination with ABCWY+OMV, ABCWY+qOMV or rMenB+OMV or MenACWY.
Time Frame: Day 1 through day 7 after any vaccination
Population: Analysis was done on the solicited safety set, ie all subjects in the all exposed set who provided postvaccination solicited AE data from day 1 (6 hours) through day 7. The all exposed set is defined as all subjects in the all enrolled population who actually received a study vaccination.
Measure: Number; unit: Participants
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB+OMV | ACWY
Number analyzed (Participants) | 108 | 110 | 115 | 99
Participants
  Injection site erythema | 57 | 53 | 72 | 30
  Injection site induration | 46 | 52 | 46 | 24
  Injection site pain | 98 | 96 | 107 | 50
  Chills | 18 | 21 | 29 | 12
  Nausea | 15 | 25 | 30 | 8
  Fatigue | 32 | 47 | 52 | 30
  Myalgia | 65 | 67 | 67 | 38
  Arthralgia | 20 | 23 | 25 | 7
  Headache | 37 | 40 | 53 | 29
  Rash | 6 | 8 | 4 | 6
  Loss of appetite | 17 | 22 | 24 | 12
  Fever ( >= 38C ) | 7 | 5 | 6 | 1
  Medically attended fever | 2 | 0 | 0 | 0
  Prophylactic use of antipyretic | 17 | 14 | 16 | 7
  Therapeutic use of antipyretic | 18 | 26 | 27 | 10

10. Secondary Outcome: The Number of Subjects Reporting Unsolicited Adverse Events After Receiving Any Vaccination in This Study.
Description: The number of subjects reporting unsolicited AEs after vaccination with ABCWY+OMV, ABCWY+qOMV, rMenB+OMV or MenACWY.
Time Frame: Throughout the study ( Day 1 to Day 241)
Population: Analysis was done on the unsolicited safety set, ie, all subjects in the all exposed set who provided postvaccination unsolicited AE data.
Measure: Number; unit: Participants
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB+OMV | ACWY
Number analyzed (Participants) | 120 | 120 | 120 | 109
Participants
  Any AEs (from day 1 to 30) | 36 | 36 | 45 | 31
  At least possibly related AEs (day 1 to 30) | 12 | 10 | 16 | 6
  Any AEs (day 31 to 60 or study termination) | 22 | 29 | 29 | 26
  At least poss.rel.AEs(day 31 to 60 or study term.) | 0 | 1 | 0 | 0
  Any AE from day 1 to 91 | 51 | 55 | 66 | 50
  At least poss.rel.AEs(day 1 to 91) | 13 | 10 | 16 | 6
  Medically attended AEs (day 92 to 241) | 26 | 24 | 30 | 31
  possibly related med.attend.AEs (day 92-241) | 0 | 0 | 0 | 0
  SAEs (Day 1 to Day 241) | 2 | 2 | 1 | 3
  Possibly/probably related SAEs | 0 | 0 | 0 | 0
  AEs leading to withdrawal (Day 1 to Day 241) | 0 | 0 | 2 | 0
  Deaths (Day 1 to Day 241) | 0 | 0 | 0 | 0

11. Post Hoc Outcome: Percentages of Subjects With hSBA Titers ≥ 1:5 Against N.Meningitidis Serogroup B Strains 44/76 and 5/99
Description: Percentages of Subjects With hSBA Titers ≥ 1:5 Against N.Meningitidis Serogroup B strains 44/76 and 5/99 at one month after second vaccination are calculated
Time Frame: At baseline and one month after second vaccination (Day 91)
Population: Analysis was done on the per-protocol population, immunogenicity. This exploratory analysis was performed only on strains 44/76 and 5/99.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB +OMV
Number analyzed (Participants) | 89 | 85 | 92
Percentage of subjects
  44/76- Baseline | 6 [2 to 12] | 7 [3 to 15] | 7 [2 to 14]
  44/76- 1 month after second dose | 100 [96 to 100] | 99 [94 to 100] | 98 [92 to 100]
  5/99- Baseline | 11 [6 to 20] | 15 [8 to 25] | 16 [9 to 25]
  5/99- 1 month after second dose | 99 [94 to 100] | 99 [94 to 100] | 98 [92 to 100]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1to Day 7; unsolicited AEs and SAEs were collected throughout the study period (Day 1 to Day 241).
Groups:
- ABCWY+OMV: Subjects in this group received two doses of rMenB(+ OMV_full dose) and MenACWY combination vaccine, administered two months apart.
- ABCWY+qOMV: Subjects in this group received two doses of rMenB (+ OMV_1/4th dose)
  +and MenACWY combination vaccine, administered two months apart.
- ACWY: Subjects in this group received first dose of placebo followed by one dose of MenACWY vaccine administered two months apart.
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB +OMV | ACWY
Serious Adverse Events (participants affected / at risk) | 2/120 | 2/120 | 1/120 | 3/109
Other Adverse Events (participants affected / at risk) | 104/120 | 104/120 | 111/120 | 87/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABCWY+OMV (N=120) | ABCWY+qOMV (N=120) | rMenB +OMV (N=120) | ACWY (N=109)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0
PERTUSSIS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 1 | 0 | 0
SPERMATOCELE (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABCWY+OMV (N=120) | ABCWY+qOMV (N=120) | rMenB +OMV (N=120) | ACWY (N=109)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 2 | 6
Nausea (Gastrointestinal disorders) | 15 | 25 | 31 | 9
Chills (General disorders) | 19 | 22 | 29 | 12
Fatigue (General disorders) | 33 | 47 | 52 | 32
Injection site Erythema (General disorders) | 59 | 53 | 72 | 32
Injection site Induration (General disorders) | 47 | 52 | 46 | 25
Injection site Pain (General disorders) | 100 | 97 | 107 | 56
Pyrexia (General disorders) | 14 | 8 | 7 | 7
Nasopharyngitis (Infections and infestations) | 3 | 8 | 6 | 5
Otitis media acute (Infections and infestations) | 2 | 0 | 2 | 6
Pharyngitis (Infections and infestations) | 7 | 8 | 7 | 5
Pharyngitis streptococcal (Infections and infestations) | 4 | 5 | 1 | 9
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 11 | 8
Decreased appetite (Metabolism and nutrition disorders) | 17 | 22 | 24 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 24 | 25 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 65 | 67 | 67 | 39
Headache (Nervous system disorders) | 38 | 41 | 53 | 32
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 6 | 9 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days